CLINICAL TRIAL: NCT06061926
Title: Effect of Celery Seed (Apium Graveolens L.) Administration on the Components of Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion
Brief Title: Effect of Celery Seed on the Components of Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Karina Griselda Pérez Rubio, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Celery Seed-MS
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome
Keywords: Celery seed; Metabolic Syndrome; Insulin resistance; Insulin secretion; Insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Double-blind, controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: Randomized double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celery seed (Experimental): 14 patients to receive homologated intervention capsule (celery seed 150 mg) one capsule with 75 mg of celery seed, every 12 hours (before breakfast and before dinner) along 12 weeks.
  Interventions: Drug: Celery Seed
- Placebo (Placebo Comparator): 14 patients to receive homologated placebo capsule (calcinated magnesia) one capsule with calcinated magnesia, every 12 hours (before breakfast and before dinner) along 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celery Seed — Celery seed capsules (Apium graveolens L.) 150 mg twice times at day, one capsule with 75 mg before breakfast and one capsule with 75 mg before dinner during 12 weeks. Homologated to the other intervention. Oral administration.
  Other Names: Apium graveolens Leen
  Arms: Celery seed
Drug: Placebo — Placebo capsules (calcined magnesia) twice times at day, one capsule before breakfast and one capsule before dinner during 12 weeks. Homologated to the other intervention. Oral administration.
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
The Metabolic Syndrome (MS) is a cluster of cardiometabolic risk factors, which include abdominal obesity, hyperglycemia, dyslipidemia, and high blood pressure. MS is a global health problem, it represents a risk factor for the progression of cardiovascular disease, which constitute the main cause of mortality in the world and in Mexico. The current treatment involves lifestyle changes and pharmacological treatment for each of the components of MS, however, there is no single approved treatment to control all components. Celery seed (Apium graveolens L.) from the Apiaceae family contains the flavonoids apigenin and luteolin; essential oils such as d-limonene, selinene and phthalides such as 3-n-butylphthalide. Thanks to its bioactive components, celery seed has proven to be effective in treating individual MS disorders; however, most studies are in animal models and there are no clinical studies that evaluate its effectiveness on all components of the system. MS, insulin sensitivity and insulin secretion so it could appear as a new, safe and effective complementary therapy for the treatment of MS.

The aim of this study is to evaluate the effect of celery seed on the components of metabolic syndrome, insulin sensitivity, and insulin secretion.

DETAILED DESCRIPTION:
A randomized, double-blind controlled clinical trial in 28 patients between 30 to 60 years of age with a diagnosis of MS according to the International Diabetes Federation (IDF) criteria without treatment and whether they voluntary accept participating and signing the informed consent.

Patients with one or more of the following criteria will be excluded: History of kidney, thyroid or liver disease; systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg, fasting glucose ≥ 126 mg/dL, triglycerides ≥ 500 mg/dL, total cholesterol ≥240 mg/dL; pregnancy or lactation; consumption of medications or supplements with effects on the study variables.

Patients included, may be withdrawn from the study if they meet any of the following conditions: Withdrawal of the informed consent, treatment adherence <80%, severe adverse reaction, intolerance or hypersensitivity to celery seed or placebo.

They will be assigned randomly two groups of 14 patients; one of the groups will receive 75 mg of celery seed twice at day (before breakfast and dinner) for 12 weeks.

The other group will receive homologated placebo (calcined magnesia) twice at day (before breakfast and dinner) for 12 weeks.

Waist circumference, blood pressure, fasting blood glucose, serum triglycerides and serum HDL cholesterol will be evaluated before and after intervention in both groups. Insulin sensitivity (Matsuda index), total insulin secretion (it is the result of the ratio between the area under the curve (AUC) of insulin in a 2-h OGTT and the AUC of glucose in a 2-h OGTT) and First phase of insulin secretion (Stumvoll index), will be calculated from the concentration of glucose and insulin obtained from an Oral Glucose Tolerance Test.

This protocol It´s already approved by the local ethics committee and written informed consent it´s going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency and dispersion, mean and deviation standard for quantitative variables; frequencies and percentage for qualitative variable. The analysis between groups (independent samples) will be analyzed using the Mann-Whitney U test for quantitative variables and the X2 test or Fisher's exact test for qualitative variables. The intragroup analysis (two related samples) will be performed using the Wilcoxon range test for quantitative variables. Statistical significance will be considered with a p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 30 and 60 years
* Diagnosis of metabolic syndrome (MS) according to the IDF criteria: waist circumference: ≥80 cm (women) ≥90 cm (men), plus two or more of the following:

  * Fasting glucose ≥ 100 mg/dL
  * Triglycerides ≥150 mg/dL
  * HDL-c: Men ≤40 mg/dL, women ≤50 mg/dL
  * Blood pressure ≥130/85 mmHg
* Body Mass Index from 25 to 34.9 kg/m²
* Stable weight at least the previous last 3 months (weight variation less than 10%)
* No pharmacological treatment for MS, insulin sensitivity and insulin secretion
* Acceptance and signing of informed consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* Glucose ≥126 mg/dL
* Total cholesterol ≥240 mg/dL
* Triglycerides ≥500mg/dL
* Systolic blood pressure ≥140 mmHg
* Diastolic blood pressure ≥90 mmHg
* Drugs or supplements consumption with proven properties that modify the behavior of the study variables.
* History of kidney, liver or thyroid disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Waist Circumference (WC) | Baseline to week 12 (end of intervention)
  Waist Circumference will be evaluated at baseline and week 12 by World Health Organization technique
Systolic Blood Pressure (SBP) | Baseline to week 12 (end of intervention)
  Systolic Blood Pressure (SBP) will be measured at baseline and week 12 with a digital sphygmomanometer three times in each arm to get an average
Diastolic Blood Pressure (DBP) | Baseline to week 12 (end of intervention)
  Diastolic Blood Pressure (DBP) will be measured at baseline and week 12 with a digital sphygmomanometer three times in each arm to get an average
High-Density Lipoprotein (HDL-c) | Baseline to week 12 (end of intervention)
  High density lipoprotein (HDL-c) level will be evaluated at baseline and week 12 by enzymatic- colorimetric technique to get c-HDL level
Fasting Blood Triglycerides Concentration (TG) | Baseline to week 12 (end of intervention)
  Fasting Blood Triglycerides Concentration (TG) level will be evaluated at baseline and week 12 by enzymatic- colorimetric technique to get triglycerides concentration
Fasting Serum Glucose (FSG) | Baseline to week 12 (end of intervention)
  The Fasting Serum Glucose (FSG) levels will be evaluated at baseline and week 12 by enzymatic- colorimetric technique to get fasting glucose level
Insulin Sensitivity (Matsuda Index) | Baseline to week 12 (end of intervention)
  Insulin sensitivity will be calculated at baseline and week 12 with Matsuda index to get insulin sensitivity
Total Insulin Secretion | Baseline to week 12 (end of intervention)
  Total insulin secretion will be calculated at baseline and week 12. It is the result of the ratio between the AUC of insulin in a 2-h OGTT and the AUC of glucose in a 2-h OGTT. It allows estimating the proportion of total insulin secretion in relation to plasma glucose concentration.
First Phase of Insulin Secretion (Stumvoll Index) | Baseline to week 12 (end of intervention)
  The first phase if insulin secretion will be calculated at baseline and week 12 with Stumvoll index to get first phase of insulin secretion

SECONDARY OUTCOMES:
Body weight | Baseline to week 12 (end of intervention)
  Body weight will be measured at baseline and week 12 with a bioimpedance analysis
Body Mass Index (BMI) | Baseline to week 12 (end of intervention)
  Body Mass Index (BMI) will be calculated at baseline and week 12 with the Quetelet index formula
Body Fat Percentage | Baseline to week 12 (end of intervention)
  Body fat percentage will be measured at baseline and week 12 with a bioimpedance analysis
Total Cholesterol (TC) | Baseline to week 12 (end of intervention)
  Total Cholesterol (TC) level will be evaluated at baseline and week 12 by enzymatic- colorimetric technique to get total cholesterol level
Low Density Lipoprotein (LDL-c) | Baseline to week 12 (end of intervention)
  Low Density Lipoprotein (LDL-c) level will be calculated at baseline and week 12 with Friedewald formula to get LDL-c level
Very Low Density Lipoprotein (VLDL) | Baseline to week 12 (end of intervention)
  Very Low Density Lipoprotein (VLDL) level will be calculated at baseline and week 12 with triglycerides concentration/5 formula to get VLDL level
Concentration of Blood Aspartate Aminostransferase (AST) | Baseline to week 12 (end of intervention)
  Concentration of Blood Aspartate Aminostransferase (AST) level will be evaluated at baseline and week 12 by enzymatic-colorimetric technique to get AST level
Alanine Aminotransferase (ALT) | Baseline to week 12 (end of intervention)
  Concentration of Blood Alanine Aminostransferase (ALT) level will be evaluated at baseline and week 12 by enzymatic-colorimetric technique to get ALT level
Creatinine | Baseline to week 12 (end of intervention)
  Concentration of creatinine level will be evaluated at baseline and week 12 by enzymatic-colorimetric technique to get creatinine level
Uric Acid | Baseline to week 12 (end of intervention)
  Concentration of uric acid level will be evaluated at baseline and week 12 by enzymatic-colorimetric technique to get uric acid level
Incidence of treatment-Emergent Adverse Events | Baseline to week 12 (end of intervention)
  Incidence of treatment-Emergent Adverse Events of celery seed or placebo will be identified by clinical evaluation from baseline week to week 12 with continuous surveillance
Tolerability to treatment | Baseline to week 12 (end of intervention)
  Tolerability to treatment of celery seed or placebo will be identified by clinical evaluation from baseline week to week 12 with continuous surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Karina G Pérez Rubio, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- INSTITUTO DE TERAPÉUTICA EXPERIMENTAL Y CLÍNICA. Centro Universitario de Ciencias de la Salud, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Escobedo-Gutierrez MJ, Cortez-Navarrete M, Martinez-Abundis E, Perez-Rubio KG. Effect of Celery Seed (Apium graveolens L.) Administration on the Components of Metabolic Syndrome, Insulin Sensitivity, and Insulin Secretion: A Clinical Trial. Pharmaceuticals (Basel). 2026 Jan 7;19(1):110. doi: 10.3390/ph19010110. PMID 41599709